## **Cover letter**

# Study title:

EUS-guided FNA with rapid on-site evaluation (ROSE) of cytopathology vs. EUS-guided FNB alone in the diagnosis of pancreatic solid lesions: a randomized controlled trial

Date of the document: 3rd of Feb 2018





## INFORMATION AND CONSENT FORM

Research Study Title: EUS-guided FNA with rapid on-site evaluation (ROSE) of

cytopathology vs. EUS-guided FNB alone in the diagnosis of pancreatic solid lesions: a randomized

controlled trial

Protocol number: 22125

**Researcher responsible for the** Yen-I Chen, MD

research study: Division of

Division of Gastroenterology and Hepatology, McGill

University Health Center, Montreal, QC, Canada

**Co-Investigator(s)/sites:** Alan Barkun, MD<sup>1</sup>

George Zogopoulos, MD<sup>2</sup>

1) Division of Gastroenterology and Hepatology, McGill University Health Center, McGill University, Montreal, QC,

Canada

2) Department of surgery, McGill University Health Center,

McGill University, Montreal, QC, Canada

Sponsor: None

#### INTRODUCTION

We are inviting you to take part in this research study because you were found to have a possible pancreatic solid mass on previous radiological tests, which will need a biopsy in order to determine the diagnosis. Possible diagnosis including a benign inflammatory mass, malignant tumor (cancer), or lymphoma.

However, before you accept to take part in this study and sign this information and consent form,

please take the time to read, understand and carefully examine the following information. You may also want to discuss this study with your family doctor, a family member or a close friend.

This form may contain words that you do not understand. We invite you to speak to the researcher responsible for this study (the "study doctor") or to other members of the research team, and ask them to explain to you any word or information that is unclear to you before you sign this form.

## **BACKGROUND**

Currently, the best way to evaluate pancreatic masses is through endoscopic-guided needle sampling of the mass to determine the diagnosis by looking at the acquired tissue under a microscope. This is done by inserting a small camera (endoscope) through the mouth of the patient then advanced to the stomach and using ultrasound guidance a sample of the pancreas can be acquired through the stomach. The sampling is usually done with a small needle called fine needle aspiration needle or FNA. FNA alone is sometimes limited due to inadequate acquisition of cells for proper diagnosis under the microscope, which can lead to need for repeat endoscopic procedures and delay in diagnosis and possibly treatment. Rapid on-site evaluation of cytopathology (ROSE) is where a cytopathologist is next to the physician doing the endoscopic procedures and evaluates each sampling performed immediately under the microscope and can give feedback to the endoscopist until enough cells has been acquired for a diagnosis. This method has been shown to increase the ability to diagnose pancreatic cancer but is expensive and requires significant amount of resources. New needles called core needles (fine needle biopsy, FNB) have recently been developed which not only acquires cells but also the entire tissue structure (histology) and has been shown to be also very accurate in the diagnosis of pancreatic cancer.

### PURPOSE OF THE RESEARCH STUDY

The purpose of this study is to compare endoscopy-guided biopsy of pancreatic masses with the new core needle (FNB), which can obtain more tissue for diagnosis vs. using a traditional needle (FNA) with the help of an immediate assessment of the obtained samples under the microscope to determine whether enough tissue has been obtained (ROSE). Both approaches have been shown to increase the accuracy of diagnosis in solid pancreatic masses but it is unclear which one is superior. This is a randomized trial meaning that you would either undergo biopsy with the new needle or with the traditional needle plus the addition of on-site assessment of the obtained samples. The advantage of the new needle is that it is easy to implement and likely much cheaper. If we can show in our study that the new needles are as accurate as FNA with ROSE then FNB could be implemented across hospitals worldwide in an easier and less expensive fashion.

For this research study, we will recruit 238 participants, men and women, ages 18 years and above. We anticipate 125 patients to be recruited at the McGill University Health Center.

#### **DESCRIPTION OF THE RESEARCH PROCEDURES**

This research study will take place at the McGill University Health Centre in including the Royal Victoria

Hospital and Montreal General Hospital. Other centers involved in this study are the Jewish General Hospital and St-Michael's Hospital (University of Toronto).

#### 1. Duration and number of visits

Your participation in this research project will last 6 months and will include 1 telephone interview following the initial procedure. The telephone interview will be approximately 5 minutes.

## 2. Study Procedure

When participating in this research project, you will be assigned to one of the following groups:

Group 1: Endoscopic ultrasound guided biopsy of the pancreas with the traditional fine needle aspirate needle with the addition of rapid on-site cytopathology (cytopathologist looking at each biopsy samples as they are taken)

Group 2: Endoscopic ultrasound guided biopsy with a novel core biopsy needle without on-site cytopathology

Furthermore, this study is randomized which means that you will be assigned to one of the groups. You may not choose the group to which you will be assigned; this process is done randomly like flipping a coin. One person out of 2 (50%) will undergo biopsy with the new needle whereas one person out of 1 (50%) will undergo biopsy with a traditional needle with the addition of rapid on-site cytopathology evaluation.

This is a single blind study, which means that you will not know which study procedure you will receive during this project. However, the study doctor will have access to this information.

## 3. Tests and procedures

During your participation in this research study, the study doctor or a member of the research team will conduct the following tests and procedures:

| DESCRIPTION OF STUDY PROCEDURES | |
|---|---|
| Procedure | Description |
| Endoscopic ultrasound guided biopsy of the pancreas | Standard of care. Whether you are part of the study or not, EUS guided biopsy of your pancreas will be recommended to you for the diagnosis of the solid mass on your pancreas. The only difference is that by being part of the study you would undergo biopsy with a novel core biopsy needle or a regular fine needle aspirate with rapid on-site evaluation of cytology of acquired samples. If you do not wish to participate in the study then you would undergo EUS-guided biopsy with a traditional fine needle aspirate alone. |

The schedule of procedures for each visit is listed below:

| SCHEDULE OF STUDY PROCEDURES | | |
|------------------------------|--------------------|--------------------|
| Procedure | Visit 1<br>(Day-0) | Visit 2<br>(Day-3) |
| EUS-guided biopsy | X | , , , |
| Telephone interview (5 min) | | Х |

## **Telephone interview:**

You will receive a phone call by one of the investigators 3 days following the procedure. We will ask you a pre-set questionnaire that will take about 5 minutes to complete. The following are the questions, which will be asked to you.

- 1) Did you experience any abdominal pain since the procedure needing medical attention? If medical intervention was required please specify:
- -Visit to the emergency room
- -Visit to an outpatient clinic
- -If inpatient, requirement for medication or increase in medication for pain control
- 2) Did you experience symptoms of nausea or vomiting?
- 3) Did you experience any bleeding needing medical attention?
- 4) Did you have any fever Temperature > 38.2 Celsius?
- 5) Any other symptoms? Please describe:

#### BENEFITS ASSOCIATED WITH THE RESEARCH STUDY

You may or may not personally benefit from your participation in this research project. However, we hope that the study results will contribute to the advancement of scientific knowledge in this field and help us find better treatments for patients.

#### RISKS ASSOCIATED WITH THE RESEARCH STUDY

The risks associated with being part of this study is best classified as minimal risks. We do not anticipate any additional risks to you by being part of the study. All associated risks are part of standard of care and standard risks associated with EUS-guided biopsy of the pancreas. Both the novel core needles and traditional fine needle aspiration with rapid on-site evaluation of cytology are part of standard of care and are not experimental.

However, if you have noticed side effects, whatever they may be, during this research study, you must tell the study doctor immediately, regardless of whether you think these effects are related to the procedure or not. Even once your participation in the study is over, do not hesitate to contact the study doctor if you experience a side effect that may be linked to the procedure.

The study doctor and members of his or her team will answer any questions that you may have regarding the risks, discomforts and side effect associated with this study. Also, at each visit, the study doctor and members of his or her team will ask you questions about any side effects you may have experienced.

#### RISKS ASSOCIATED WITH PREGNANCY

If you are pregnant you will not be a candidate for the study.

#### **VOLUNTARY PARTICIPATION AND THE RIGHT TO WITHDRAW**

Your participation in this research project is voluntary. Therefore, you may refuse to participate. You may also withdraw from the project at any time, without giving any reason, by informing the study doctor or a member of the research team.

Your decision not to participate in the study, or to withdraw from it, will have no impact on the quality of care and services to which you are otherwise entitled, or on your relationship with the study doctor or clinical team.

The study doctor, the Research Ethics Board, the funding agency, or the Sponsor may put an end to your participation without your consent. This may happen if new findings or information indicate that participation is no longer in your interest, if you do not follow study instructions, or if there are administrative reasons to terminate the project.

If you withdraw or are withdrawn from the study, the information and biological material already collected for the study will be stored, analyzed and used to ensure the integrity of the study.

Any new findings that could influence your decision to stay in the research project will be shared with you as soon as possible.

## CONFIDENTIALITY

During your participation in this study, the study doctor and their team will collect and record information about you in a study file. They will only collect information required to meet the scientific goals of the study.

The study file may include information from your medical chart, including your identity, concerning your past and present state of health, your lifestyle, as well as the results of the tests, exams, and procedures that you will undergo during this research project. Your research file could also contain other information, such as your name, sex, date of birth and ethnic origin.

No tissue samples will be acquired for research purposes. All collected samples during EUS-guided biopsy will be received by the cytopathology lab and stored as per standard practice of the institution.

All the information collected during the research project will remain strictly confidential to the extent provided by law. You will only be identified by a code number. The key to the code linking your name to your study file will be kept by the study doctor.

To ensure your safety, a copy of this information and consent form be placed in your medical chart. As

a result, any person or company to whom you give access to your medical chart will have access to this information.

The study data will be stored for 25 years by the study doctor.

The data may be published or shared during scientific meetings; however it will not be possible to identify you.

For monitoring, control, safety, security, and marketing of a new study drug, your study file as well as your medical charts may be examined by a person mandated by Canadian or international regulatory authorities, such as Health Canada, as well as by representatives of the study sponsor, the institution, or the Research Ethics Board. All these individuals and organizations adhere to policies on confidentiality.

You have the right to consult your study file in order to verify the information gathered, and to have it corrected if necessary.

However, in order to protect the scientific integrity of the research project, accessing certain information before the project is ended may require that you be withdrawn from the study.

#### **INCIDENTAL FINDINGS**

Material incidental findings are findings made in the course of the study that may have significant impacts on your current or future wellbeing or that of your family members. A material incidental finding concerning you in the course of this research will be communicated to you and to a health professional of your choice.

Incidental findings often occur during any endoscopic ultrasound exam. However, the endoscopic ultrasound exam that you will undergo is standard of care. Meaning that whether you are part of this study or not, the exam will be recommended to you. Any incidental finding will therefore be treated as clinically indicated and you will be informed immediately of all findings.

#### MARKETING POSSIBILITIES

The research results, including those following your participation in this study, could lead to the creation of commercial products. However, you will not receive any financial benefits.

## **FUNDING OF THE RESEARCH PROJECT**

The study doctor and the institution have not received funding from the sponsor for the completion of the research project.

#### **COMPENSATION**

You will not receive financial compensation for participating in this research study.

#### SHOULD YOU SUFFER ANY HARM

Should you suffer harm of any kind following the endoscopic procedure, or following any other procedure related to the research study, you will receive the appropriate care and services required by your state of health.

By agreeing to participate in this research project, you are not waiving any of your legal rights nor discharging the study doctor, the sponsor or the institution, of their civil and professional responsibilities.

#### **CLINICAL TRIAL REGISTRATION**

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>. This Website will not include information that can identify you. At most, the Website will include a summary of the results. You can search this Website at any moment.

## **CONTACT INFORMATION**

If you have questions or if you have a problem you think may be related to your participation in this research study, or if you would like to withdraw, you may communicate with the study doctor or with someone on the research team at the following number: 514-934-1934 Ext: 34868.

For any question concerning your rights as a research participant taking part in this study, or if you have comments, or wish to file a complaint, you may communicate with:

The Patient Ombudsman of the McGill University Health Center at the following: 514-934-1934 Ext: 48306.

## **OVERVIEW OF ETHICAL ASPECTS OF THE RESEARCH**

The McGill University Health Centre Research Ethics Board reviewed this study and is responsible for monitoring it at all participating institutions in the health and social services network in Quebec.

| Research Study Title: | EUS-guided FNA with rapid on-site evaluation (ROSE) of cytopathology vs. EUS-guided FNB alone in the diagnosis of pancreatic solid lesions: a randomized controlled trial |
|---|---|
| SIGNATURES | |
| Signature of the participant | |
| consent form were explained to me | d consent form. Both the research study and the information and e. My questions were answered, and I was given sufficient time to consent to participate in this research study in accordance with the |
| I authorize the research study team | to have access to my medical record for the purposes of this study. |
| Name of participant | Signature Date |
| Signature of the person obtaining of | onsent |
| I have explained the research study participant, and I answered all his/ho | and the terms of this information and consent form to the research er questions. |
| Name of the person obtaining conse | ent Signature Date |
| Commitment of the principal invest | igator |
| I certify that this information and continuous the questions the participant had we | consent form were explained to the research participant, and that ere answered. |
| = | arch team, to respect what was agreed upon in the information and nd nd dated copy of this form to the research participant. |

Name of the principal investigator

Signature

Date